CLINICAL TRIAL: NCT03462498
Title: Study to Evaluate the Safety of Reducing Dual Antiplatelet Therapy (DAPT) Duration to 1 Month for Patients With Acute Coronary Syndrome (ACS) After Implantation of Everolimus-eluting Cobalt-chromium Stent
Brief Title: ShorT and OPtimal Duration of Dual AntiPlatelet Therapy-2 Study for the Patients With ACS
Acronym: STOPDAPT-2 ACS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Takeshi Morimoto, Professor of Medicine, Kyoto University, Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C1348
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Acute Coronary Syndrome; Acute Myocardial Infarction; Coronary Artery Disease; Percutaneous Coronary Intervention; Platelet Aggregation Inhibitors
Keywords: Acute Coronary Syndrome; Acute Myocardial Infarction; Coronary Artery Disease; Percutaneous Coronary Intervention; Platelet Aggregation Inhibitors
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-month DAPT (Active Comparator): 1-month dual antiplatelet therapy (DAPT) composed of aspirin and P2Y12 receptor antagonists and clopidogrel monotherapy for 59 months
  Interventions: Drug: 1-months DAPT
- 12-month DAPT (Active Comparator): 1-month dual antiplatelet therapy (DAPT) composed of aspirin and P2Y12 receptor antagonists; 11-month DAPT composed of aspirin and clopidogrel and aspirin monotherapy for 48 months
  Interventions: Drug: 12-month DAPT

INTERVENTIONS:
Drug: 1-months DAPT — 1-month DAPT followed by 59-month monotherapy
  Arms: 1-month DAPT
Drug: 12-month DAPT — 12-month DAPT followed by 48-month monotherapy
  Arms: 12-month DAPT

SUMMARY:
The purpose of this study is to evaluate the safety of reducing dual antiplatelet therapy (DAPT) duration to 1 month after implantation of the everolimus-eluting cobalt-chromium stent (CoCr-EES) under the setting of acute coronary syndrome (ACS).

DETAILED DESCRIPTION:
The drug-eluting stents (DESs) are currently used in the majority of percutaneous coronary intervention (PCI) procedures. On the other hand, the problems of the first-generation DES (late adverse events, such as very late stent thrombosis) have been pointed out. Dual antiplatelet therapy (DAPT) has become a standard regimen after DES implantation and for fear of very late stent thrombosis, DAPT is frequently performed for 1 year or longer in clinical practice. Especially guidelines recommend 1-year DAPT for patients with acute coronary syndrome (ACS), though its rational is based on the study more than 15 years old. However, serious hemorrhagic complications associated with prolonged DAPT duration can bring disadvantages to patients, and it is extremely important to clarify an optimal DAPT duration after DES procedure. Currently, 1-month DAPT regimen after bare metal stent (BMS) implantation is commonly used in clinical practice, producing no major problems. Based on a meta-analysis of recent clinical studies, it has also been reported that the use of Cobalt-Chromium Everolimus-Eluting Stent (CoCr-EES) reduces the risk of early stent thrombosis by half compared to the use of BMS. There is no necessity to extend antiplatelet therapy after CoCr-EES implantation longer than after BMS implantation, and it is considered possible to use the same 1-month DAPT duration as after BMS implantation. The investigators already planned and started a multicenter, randomized, open-label, controlled study, in which the subjects who have undergone CoCr-EES procedure will be divided into the 1-month DAPT and clopidogrel monotherapy group and the 12-month DAPT and aspirin monotherapy group (STOPDAPT-2; NCT02619760), where primary endpoint is the incidence of composite events including cardiovascular death, myocardial infarction, stent thrombosis, stroke, and bleeding defined by TIMI major or minor bleeding. In STOPDAPT-2, the non-inferiority about primary endpoint of 1-month DAPT group will be evaluated at 12 months after index procedure and secondarily, the superiority about primary endpoint of 1-month DAPT group will be evaluated at 5 years after index procedure. The proportion of patients with ACS is about 30-40% in STOPDAPT-2 and the power is insufficient to evaluate the safety and efficacy of 1-month DAPT regimen specifically for patients with ACS. Therefore the investigators planned the current study to enroll patients of ACS with the same protocol as STOPDAPT-2.

ELIGIBILITY:
Inclusion Criteria:

* Patients received percutaneous coronary intervention with cobalt-chromium everolimus-eluting stent under the setting of acute coronary syndrome
* Patients who are capable of oral dual antiplatelet therapy consisting of aspirin and P2Y12 receptor antagonist

Exclusion Criteria:

* Patients requiring oral anticoagulants
* Patients with medical history of intracranial hemorrhage
* Patients who have experienced serious complications (myocardial infarction, stroke, and major bleeding) during hospital stay after percutaneous coronary intervention
* Patients with drug eluting stents other than Cobalt chromium everolimus eluting stents implanted at the time of enrollment
* Patients confirmed to have no tolerability to clopidogrel before enrollment
* Patients requiring continuous administration of antiplatelet drugs other than aspirin and P2Y12 receptor antagonists at the time of enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3008 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Composite event of cardiovascular death/myocardial infarction/definite stent thrombosis/stroke/bleeding defined as major or minor under the definition of Thrombolysis in Myocardial Infarction (TIMI) Study group | 12 months
Composite event of cardiovascular death/myocardial infarction/definite stent thrombosis/stroke/bleeding defined as major or minor under the definition of Thrombolysis in Myocardial Infarction (TIMI) Study group | 60 months

SECONDARY OUTCOMES:
Composite event of cardiovascular death/myocardial infarction/definite stent thrombosis/stroke | 12 months
Composite event of cardiovascular death/myocardial infarction/definite stent thrombosis/stroke | 60 months
Bleeding defined as major or minor under the definition of Thrombolysis in Myocardial Infarction (TIMI) Study group | 12 months
Bleeding defined as major or minor under the definition of Thrombolysis in Myocardial Infarction (TIMI) Study group | 60 months
Upper gastrointestinal endoscopic examination or treatment | 60 months
Composite event of all-cause death/myocardial infarction | 12 months
Composite event of all-cause death/myocardial infarction | 60 months
All-cause death | 12 months
All-cause death | 60 months
Composite event of cardiovascular death/myocardial infarction | 12 months
Composite event of cardiovascular death/myocardial infarction | 60 months
Cardiovascular death | 12 months
Cardiovascular death | 60 months
Myocardial infarction | 12 months
Myocardial infarction | 60 months
Stroke | 12 months
Stroke | 60 months
Definite stent thrombosis | 12 months
  Academic Research Consortium definition
Definite stent thrombosis | 60 months
  Academic Research Consortium definition
Target lesion failure | 12 months
Target lesion failure | 60 months
Target vessel failure | 12 months
Target vessel failure | 60 months
Major adverse cardiac event | 12 months
  Composite of cardiac death, myocardial infarction, and clinically-driven TLR
Major adverse cardiac event | 60 months
  Composite of cardiac death, myocardial infarction, and clinically-driven TLR
Target lesion revascularization | 12 months
Target lesion revascularization | 60 months
Clinically-driven target lesion revascularization | 12 months
Clinically-driven target lesion revascularization | 60 months
Non target lesion revascularization | 12 months
Non target lesion revascularization | 60 months
Coronary artery bypass graft | 12 months
Coronary artery bypass graft | 60 months
Target vessel revascularization | 12 months
Target vessel revascularization | 60 months
Any coronary revascularization | 12 months
Any coronary revascularization | 60 months
Bleeding complications | 12 months
Bleeding complications | 60 months
Gastrointestinal bleeding | 12 months
Gastrointestinal bleeding | 60 months
Gastrointestinal complaints requiring upper gastrointestinal endoscopy | 12 months
Gastrointestinal complaints requiring upper gastrointestinal endoscopy | 60 months
Newly diagnosed cancer | 60 months
  The endpoint is a newly diagnosed malignancy during the follow-up period that has not been previously diagnosed before enrollment. This does not include recurrent tumor after remission, includes early-stage cancer eligible for endoscopic treatment, and includes the tumors which are not diagnosed by tissue biopsy but are judged to be clinically malignant on imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Takeshi Kimura, MD, Principal Investigator — Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine
Locations (1):
- Kyoto University Graduate School of Medicine, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yamamoto K, Watanabe H, Morimoto T, Obayashi Y, Natsuaki M, Domei T, Yamaji K, Suwa S, Isawa T, Watanabe H, Yoshida R, Sakamoto H, Akao M, Hata Y, Morishima I, Tokuyama H, Yagi M, Suzuki H, Wakabayashi K, Suematsu N, Inada T, Tamura T, Okayama H, Abe M, Kawai K, Nakao K, Ando K, Tanabe K, Ikari Y, Morino Y, Kadota K, Furukawa Y, Nakagawa Y, Kimura T; STOPDAPT-2 and STOPDAPT-2 ACS Investigators. Clopidogrel Monotherapy After 1-Month DAPT in Patients With High Bleeding Risk or Complex PCI. JACC Asia. 2023 Jan 10;3(1):31-46. doi: 10.1016/j.jacasi.2022.09.011. eCollection 2023 Feb. PMID 36873770
- [Derived] Yamamoto K, Watanabe H, Morimoto T, Obayashi Y, Natsuaki M, Yamaji K, Domei T, Ogita M, Ohya M, Tatsushima S, Suzuki H, Tada T, Ishii M, Nikaido A, Watanabe N, Fujii S, Mori H, Nishikura T, Suematsu N, Hayashi F, Komiyama K, Shigematsu T, Isawa T, Suwa S, Ando K, Kimura T; STOPDAPT-2 and STOPDAPT-2 ACS Investigators. Clopidogrel Monotherapy After 1-Month Dual Antiplatelet Therapy in Patients With Diabetes Undergoing Percutaneous Coronary Intervention. JACC Cardiovasc Interv. 2023 Jan 9;16(1):19-31. doi: 10.1016/j.jcin.2022.09.053. Epub 2022 Dec 14. PMID 36599584
- [Derived] Obayashi Y, Watanabe H, Morimoto T, Yamamoto K, Natsuaki M, Domei T, Yamaji K, Suwa S, Isawa T, Watanabe H, Yoshida R, Sakamoto H, Akao M, Hata Y, Morishima I, Tokuyama H, Yagi M, Suzuki H, Wakabayashi K, Suematsu N, Inada T, Tamura T, Okayama H, Abe M, Kawai K, Nakao K, Ando K, Tanabe K, Ikari Y, Morino Y, Kadota K, Furukawa Y, Nakagawa Y, Kimura T; STOPDAPT-2 and STOPDAPT-2 ACS Investigators. Clopidogrel Monotherapy After 1-Month Dual Antiplatelet Therapy in Percutaneous Coronary Intervention: From the STOPDAPT-2 Total Cohort. Circ Cardiovasc Interv. 2022 Aug;15(8):e012004. doi: 10.1161/CIRCINTERVENTIONS.122.012004. Epub 2022 Aug 1. PMID 35912647
- [Derived] Watanabe H, Morimoto T, Natsuaki M, Yamamoto K, Obayashi Y, Ogita M, Suwa S, Isawa T, Domei T, Yamaji K, Tatsushima S, Watanabe H, Ohya M, Tokuyama H, Tada T, Sakamoto H, Mori H, Suzuki H, Nishikura T, Wakabayashi K, Hibi K, Abe M, Kawai K, Nakao K, Ando K, Tanabe K, Ikari Y, Morino Y, Kadota K, Furukawa Y, Nakagawa Y, Kimura T; STOPDAPT-2 ACS Investigators. Comparison of Clopidogrel Monotherapy After 1 to 2 Months of Dual Antiplatelet Therapy With 12 Months of Dual Antiplatelet Therapy in Patients With Acute Coronary Syndrome: The STOPDAPT-2 ACS Randomized Clinical Trial. JAMA Cardiol. 2022 Apr 1;7(4):407-417. doi: 10.1001/jamacardio.2021.5244. PMID 35234821